CLINICAL TRIAL: NCT07222059
Title: A Phase 3, Single Arm, Open Study to Assess the Immunogenicity and Safety of vYF in Adults Aged 18 Years and Over
Brief Title: Phase 3 Single Arm, Open Study on vYF in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VYF00011; VYF00011 (Other: Sanofi Identifier)
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- vYF (Experimental): One single dose of vYF will be administered subcutaneously at the 1st visit
  Interventions: Biological: Yellow fever vaccine (live)

INTERVENTIONS:
Biological: Yellow fever vaccine (live) — Pharmaceutical form:Powder and diluent for suspension for injection-Route of administration:Subcutaneous
  Other Names: vYF vaccine

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of vYF in adults aged 18 years and over in Japan.

Study details include:

* The study duration will be up to approximately 1 month.
* One single dose of vYF will be administrated subcutaneously at the 1st visit.
* The visit frequency will be Day 01 (Visit 01) and Day 29 (Visit 02). One telephone call (TC) will be planned at Day 15.

Number of Participants:

A total of 254 participants is expected to be included in the study with the aim to obtain a total of 203 evaluable participants.

Study Arms and Duration:

Eligible participants will receive, subcutaneously, a single dose of vYF vaccine on Day 1.

The duration of each participation will be approximately 1 month for each participant.

DETAILED DESCRIPTION:
Duration of study participation: approximately 1 month for each participant

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years on the day of inclusion*

  * "From 18 years" means from the day of the 18th birthday
* Participants who are healthy as determined by medical evaluation including medical history and physical examination.
* Able to attend all scheduled visits and to comply with all study procedures
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR

. Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration.

A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) before any dose of study intervention on Day 01 and will be repeated on Day 29 to confirm the participant is still not pregnant within the 28 days of vaccine administration.

- Informed consent form (ICF) has been signed and dated Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy, or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known history or laboratory evidence of HIV infection.
* Known history of hepatitis B or hepatitis C seropositivity
* Known history of FV infection, Japanese encephalitis (JE) excluded
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Personal or family history of thymic pathology (thymoma, thymectomy, or myasthenia).
* Chronic illness* that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion, including malignancy, such as leukemia, or lymphoma

  * Chronic illness may include, but is not limited to cardiac disorders, renal disorders, auto-immune disorders, diabetes, psychiatric disorders or chronic infection
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 37.5°C [or ≥ 99.5°F]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following the study vaccination (prior to Visit 2 on Day 29), except for influenza vaccination, which may be received at least 2 weeks before study vaccines. This exception includes pandemic influenza vaccines including monovalent pandemic influenza vaccines.
* Previous vaccination against YF.
* Receipt of immune globulins, blood, or blood-derived products in the past 6 months.
* Administration of any anti-viral within 2 months preceding the vaccination and up to the 6 weeks following the vaccination.
* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the course of the study in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Planned travel in a YF endemic country within 28 days of investigational vaccine administration.
* For participants greater than 60 years at the time of enrolment: any underlying medical condition (eg, cardiovascular disorders, organ failure) which could increase risk of a serious viscerotropic event or serious neurologic events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2025-10-23 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with seroconversion to YF virus in YF-naive participants | 28 days after one dose of vYF vaccine
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in neutralizing Ab (NAb) titers as compared to the pre-vaccination value (Day 01)

SECONDARY OUTCOMES:
Percentage of participants with seroprotection to YF virus | At Day 01 and Day 29
  Seroprotection is defined as NAb titers ≥ 10 (1/dil) at the corresponding timepoint
Percentage of participants with seroconversion to YF virus | 28 days after one dose of vYF vaccine
  Seroconversion rates will be assessed using a YF MN assay Seroconversion is defined as a 4-fold increase in neutralizing Ab (NAb) titers as compared to the pre-vaccination value (Day 01)
Geometric Mean Titers (GMTs) of neutralizing antibodies against YF virus | At Day 01 and Day 29
  Antibody titers are expressed as GMTs
Geometric Mean Titers Ratio (GMTRs) of neutralizing antibodies against YF virus | At Day 01 and Day 29
  GMTRs Day 29/Day 01
Number of participants with immediate adverse events | Within 30 minutes after vaccination
  Immediate adverse events are any unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site reactions | Within 7 days after vaccination
  Solicited injection site reactions: injection site pain, injection site erythema, injection site swelling
Number of participants with solicited systemic reactions | Within 14 days after vaccination
  Solicited systemic reactions: fever, headache, fatigue, myalgia
Number of participants with unsolicited adverse events (AEs), including adverse events of special interest (AESIs) | Within 28 days after vaccination
  Unsolicited (spontaneously reported) AEs, not fulfilling criteria for solicited adverse reactions, including AESIs
Number of participants with serious adverse events (SAEs) including serious AESIs | Within 28 days after vaccination
  SAEs including serious AESIs
Number of participants with related SAEs and all deaths | From Day 01 to Day 29 after vaccination
  Related SAEs and all deaths

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Investigational Site Number : 3920001, Takatsuki, Osaka
  - Investigational Site Number : 3920002, Chūō, Tokyo
  - Investigational Site Number : 3920003, Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920004, Taitō City, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VYF00011 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26934&tenant=MT_SNY_9011